CLINICAL TRIAL: NCT04203316
Title: An Open-Label Feasibility Study to Assess the Safety and Pharmacokinetics of Enasidenib in Pediatric Patients With Relapsed/Refractory Acute Myeloid Leukemia (R/R-AML) With an Isocitrate Dehydrogenase-2 (IDH2) Mutation
Brief Title: Enasidenib for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia Patients With an IDH2 Mutation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL18P1; NCI-2019-07902 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL18P1 (Other: Children's Oncology Group); ADVL18P1 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-12-04; First posted 2019-12-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; enasidenib; 2-Propanol; methanesulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (enasidenib) (Experimental): Patients receive enasidenib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and/or biopsy and collection of blood on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Enasidenib; Drug: Enasidenib Mesylate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Enasidenib — Given PO
  Other Names: AG 221; AG-221; AG221; CC-90007 Free Base
Drug: Enasidenib Mesylate — Given PO
  Other Names: 2-Methyl-1-[(4-[6-(trifluoromethyl)pyridin-2-yl]-6-{[2-(trifluoromethyl)pyridin-4-yl]amino}-1,3,5-triazin-2-yl)amino]propan-2-ol Methanesulfonate; 2-Propanol, 2-Methyl-1-((4-(6-(trifluoromethyl)-2-pyridinyl)-6-((2-(trifluoromethyl)-4-pyridinyl)amino)-1,3,5-triazin-2-yl)amino)-, Methanesulfonate (1:1); AG-221 Mesylate; CC 90007; CC-90007; CC90007; Enasidenib Methanesulfonate; Idhifa

SUMMARY:
This phase II trial studies the side effects of enasidenib and sees how well it works in treating pediatric patients with acute myeloid leukemia that has come back after treatment (relapsed) or has been difficult to treat with chemotherapy (refractory). Patients must also have a specific genetic change, also called a mutation, in a protein called IDH2. Enasidenib may stop the growth of cancer cells by blocking the mutated IDH2 protein, which is needed for leukemia cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of treatment with enasidenib mesylate (enasidenib) administered at continuous daily oral dosing for a 28-day cycle up to 12 cycles in pediatric patients with IDH2-mutant relapsed/refractory (R/R)-acute myeloid leukemia (AML).

II. To characterize the plasma pharmacokinetic (PK) profile of enasidenib in pediatric patients with IDH2-mutant R/R-AML.

SECONDARY OBJECTIVES:

I. To investigate the pharmacodynamic (PD) relationship of oncogenic metabolite 2-hydroxyglutarate (2-HG) to enasidenib treatment in pediatric patients with IDH2-mutant R/R-AML.

II. To describe the clinical activity of enasidenib in pediatric patients with IDH2-mutant R/R-AML.

IIa. Clinical activity will be defined as:

IIai. Overall response rate (ORR) using response criteria adapted from the AML International Working Group Criteria; IIaii. Composite complete remission rate (CCRR) defined as complete remission (CR) and complete remission with incomplete blood count recovery (CRi); IIaiii. Time to response (TTR); IIaiv. Time to complete remission (TTCR); IIav. Duration of response (DOR); IIavi. Duration of CR (DOCR); IIavii. Event-free survival (EFS) and overall survival (OS).

OUTLINE:

Patients receive enasidenib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and/or biopsy and collection of blood on study.

After completion of study treatment, patients are followed up at 30 days, then periodically up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 24 months and < 21 years of age at the time of study enrollment
* Patient must have AML with an IDH2 mutation identified from a peripheral blood or bone marrow sample at the time of diagnosis and/or relapsed/refractory disease
* Patient must have bone marrow assessment (aspiration or biopsy) with > 5% leukemic blasts by morphology and/or flow cytometry in at least one of the following clinical scenarios:

  * Second or greater relapse after chemotherapy or hematopoietic stem cell transplant (HSCT)
  * Refractory after >= 2 attempts at induction therapy
* Relapsed patients

  * Must not have received prior re-induction therapy for this relapse
  * Each block of chemotherapy (i.e., cytarabine, daunorubicin and etoposide [ADE], cytarabine and mitoxantrone [MA]) is a separate re-induction attempt
  * Donor lymphocyte infusion (DLI) is considered a re-induction attempt
* Refractory patients

  * Each attempt at induction therapy may include up to two chemotherapy courses
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Evaluation of cerebrospinal fluid (CSF) is only required if there is a clinical suspicion of central nervous system (CNS) involvement by leukemia during eligibility screening. Should a patient be found to have CNS2 or CNS3 status by CSF prior to eligibility screening, patient may receive intrathecal chemotherapy > 72 hours prior to starting study drug. CNS1 status must be established before starting study drug
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g., blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment

    * >= 14 days must have elapsed after the completion of other cytotoxic therapy with the exception of hydroxyurea. Additionally, patients must have fully recovered from all acute toxic effects of prior therapy. NOTE: Cytoreduction with hydroxyurea must be discontinued >= 24 hours prior to the start of protocol therapy
    * Intrathecal chemotherapy must be completed >= 72 hours prior to the start of the first cycle of treatment
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion:

      * >= 60 days after infusion for bone marrow or stem cell transplant and
      * >= 4 weeks after infusion for any stem cell infusion including DLI or boost infusion
      * There must be no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular Therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * XRT/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-metaiodobenzylguanidine [MIBG]): >= 42 days after systemically administered radiopharmaceutical therapy
  * Study-specific limitations on prior therapy: small molecule investigational agents: >= 14 days or > 5 half-lives must have elapsed from the last dose of the agent, whichever is greater
* Platelet count >= 20,000/mm^3 (may receive platelet transfusions)
* Hemoglobin >= 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate [GFR] >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age: Maximum serum creatinine (mg/dL)

    * 2 to < 6 years: 0.8 (male and female)
    * 6 to < 10 years: 1 (male and female)
    * 10 to < 13 years: 1.2 (male and female)
    * 13 to < 16 years: 1.5 (male); 1.4 (female)
    * >= 16 years: 1.7 (male); 1.4 (female)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 225 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* Left ventricular ejection fraction of >= 50% by echocardiogram
* Regulatory Requirements

  * All patients and/or their parents or legal authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines
  * All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* AML associated with Down syndrome or t(15;17) is not eligible for study
* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study therapy and for 2 months after the last dose of enasidenib. Abstinence is an acceptable method of birth control. It is not known if enasidenib is present in breast milk. Breastfeeding is not recommended during therapy or for at least 30 days after the last dose of enasidenib
* Concomitant Medications:

  * Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid. The use of corticosteroids to manage the side effect of IDH inhibitor-associated differentiation syndrome (IDH-DS), is permitted on study
  * Investigational drugs: Patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer agents: Patients who are currently receiving other anti-cancer agents are not eligible (except leukemia patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy; the use of hydroxyurea to manage the side effect of IDH-DS, is permitted on study)
  * Anti-GVHD agents post-transplant: Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients must be able to swallow intact tablets whole or use the alternate enasidenib formulation.

  * Patients with known hypersensitivity to any of the components of enasidenib are not eligible.
  * Patients with prior exposure to enasidenib or another IDH2 inhibitor are not eligible.
  * Patients taking the following drugs will be excluded from study entry unless these drugs are discontinued or patients are transferred to a medically acceptable alternative > 5 half-lives before the first dose of enasidenib.

    * Drugs with a narrow therapeutic range that are sensitive substrates of the following cytochrome P450 (CYP) enzymes: CYP2C8 (e.g. paclitaxel), 2C9 (e.g. phenytoin and warfarin), 2C19 (e.g. s-mephenytoin), 2D6 (e.g. thioridazine), and 1A2 (e.g. theophylline and tizanidine).
    * Breast cancer resistant protein (BCRP) transporter-sensitive substrate rosuvastatin
* Patients with the following leukemia complications are not eligible for this trial:

  * No intrathecal chemotherapy is permitted on study. Prior to study enrollment, cerebrospinal fluid (CSF) evaluation is only required if there is a clinical suspicion for CNS leukemia. Clinical signs of CNS leukemia (such as facial nerve palsy, brain/eye involvement or hypothalamic syndrome) are not eligible for this trial
  * Immediately life-threatening, severe complications of leukemia including uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
* Patients who have received a prior solid organ transplantation are not eligible
* Infection: Patients who have an uncontrolled infection or patients with known human immunodeficiency virus (HIV) or active hepatitis B or C are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 24 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-10-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities of enasidenib | Up to 28 days
  Frequencies (%) of patients with cycle 1 dose limiting toxicity stratified by dose level.
Area under the plasma concentration versus time curve of enasidenib | Up to 2 days
  A descriptive analysis of the area under the plasma concentration versus time curve of enasidenib during cycle 1 at pre-dose and 1, 2, 4, 6, and 24 hours post-dose including median, minimum and maximum stratified by dose level.
Total plasma clearance of enasidenib | Up to 2 days
  A descriptive analysis of the total plasma clearance of enasidenib during cycle 1 at pre-dose and 1, 2, 4, 6, and 24 hours post-dose including median, minimum and maximum by dose level.
Elimination half-life of enasidenib | Up to 2 days
  A descriptive analysis of the elimination half-life of enasidenib during cycle 1 at pre-dose and 1, 2, 4, 6, and 24 hours post-dose including median, minimum and maximum by dose level.
Maximum concentration of enasidenib | Up to 2 days
  A descriptive analysis of the maximum concentration of enasidenib during cycle 1 at pre-dose and 1, 2, 4, 6, and 24 hours post-dose including median, minimum and maximum by dose level.

SECONDARY OUTCOMES:
Plasma 2-HG levels of enasidenib | Up to 84 days
  A descriptive analysis of the plasma 2-HG levels observed pre-dose at day 0, 28, and 84 of enasidenib including median, minimum and maximum by dose level.
Overall Response Rate of enasidenib | Up to 2 years
  Frequency (%) of patients with at least partial response by dose level.
Composite complete remission rate (complete remission [CR]/ CR with incomplete hematologic recovery [CRi]) | Up to 2 years
  Will be reported in a table as frequency of response (%) for total overall response rate (ORR) stratified by dose level.
Time to response of enasidenib | Up to 2 years
  Median time to response with 95% confidence interval stratified by dose level.
Time to complete remission of enasidenib | Up to 2 years
  Median time to remission with 95% confidence interval stratified by dose level.
Duration of response of enasidenib | Up to 2 years
  Median duration of response with minimum and maximum stratified by dose level.
Duration of complete response of enasidenib | Up to 2 years
  Median duration of remission with minimum and maximum stratified by dose level.
Event-free survival of enasidenib | Up to 2 years
  Median time to event with 95% confidence interval stratified by dose level.
Overall survival of enasidenib | Up to 2 years
  Median time to death with 95% confidence interval stratified by dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Zarnegar-Lumley, Principal Investigator — Children's Oncology Group
Locations (28):
- United States (27):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada

DOCUMENTS (1):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT04203316/Prot_000.pdf